CLINICAL TRIAL: NCT05152485
Title: A Phase 1, Randomized, Open-Label, Parallel-Arm Study to Evaluate the Relative Bioavailability of Two Formulations of BIIB104 and Assess the Effect of Food on the Pharmacokinetics of BIIB104 Following Administration of a Single, Fixed, Oral Dose of BIIB104 in Healthy Participants
Brief Title: A Study to Evaluate the Relative Bioavailability of Two Formulations of BIIB104 and Assess the Effect of Food on the Pharmacokinetics of BIIB104 Following Administration of a Single, Fixed, Oral Dose of BIIB104 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 263HV109
Record Dates: First submitted 2021-12-08; First posted 2021-12-09 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BIIB104 0.5 mg Reference Formulation (Fasted State) (Active Comparator): Participants will receive BIIB104 0.5 mg, immediate-release liquid-filled hard-shell capsule, orally, on Day 1 in the fasted state.
  Interventions: Drug: BIIB104 Reference Formulation
- BIIB104 0.5 mg Test Formulation (Fasted State) (Experimental): Participants will receive BIIB104 0.5 mg, immediate-release softgel capsule, orally, on Day 1 in the fasted state.
  Interventions: Drug: BIIB104 Test Formulation
- BIIB104 0.5 mg Test Formulation (Fed State) (Experimental): Participants will receive BIIB104 0.5 mg, immediate-release softgel capsule, orally, on Day 1 in the fed state.
  Interventions: Drug: BIIB104 Test Formulation

INTERVENTIONS:
Drug: BIIB104 Reference Formulation — Administered as specified in the treatment arm
  Arms: BIIB104 0.5 mg Reference Formulation (Fasted State)
Drug: BIIB104 Test Formulation — Administered as specified in the treatment arm
  Arms: BIIB104 0.5 mg Test Formulation (Fasted State); BIIB104 0.5 mg Test Formulation (Fed State)

SUMMARY:
The primary objectives of this study are to evaluate the relative bioavailability of the BIIB104 test formulation compared with the reference formulation in healthy Caucasian male adult participants in the fasted state and to assess the impact of food on BIIB104 pharmacokinetic (PK) parameters for the test formulation in healthy Caucasian male adult participants.

The secondary objective of the study is to assess the safety and tolerability of BIIB104 0.5 milligrams (mg) test formulation in the fasted and fed states following single-dose administration.

ELIGIBILITY:
Key Inclusion Criteria:

* Has a body mass index (BMI) between 18 and 30 kilogram per square meter (kg/m^2), inclusive and a total body weight >50 kilograms [110 pound (lb)].

Key Exclusion Criteria:

* Participates in other studies involving treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to randomization and/or during study participation.
* Previously participated in this study or previous studies with BIIB104.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve from Time Zero to Time of the Last Measurable Concentration (AUClast) of BIIB104 | Up to Day 6
Area Under the Plasma Concentration-Time Curve from Time Zero to Infinity (AUCinf) of BIIB104 | Up to Day 6
Maximum Observed Plasma Concentration (Cmax) of BIIB104 | Up to Day 6
Time to Reach Maximum Observed Plasma Concentration (Tmax) for BIIB104 | Up to Day 6

SECONDARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | From Day 1 up to end of study (up to Day 16)
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. TEAEs are AEs that start or worsen after receiving the study drug. An SAE is any untoward medical occurrence that at any dose results in death; in the view of the investigator, places the participant at immediate risk of death (a life-threatening event); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect or is a medically important event.
Number of Participants with Clinically Significant Abnormalities in Clinical Laboratory Parameters | From Day 1 up to end of study (up to Day 16)
Number of Participants with Clinically Significant Abnormalities in Vital Signs | From Day 1 up to end of study (up to Day 16)
Number of Participants with Clinically Significant Abnormalities in Physical Examination Parameters | From Day 1 up to end of study (up to Day 16)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- QPS MRA, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/